CLINICAL TRIAL: NCT03396198
Title: An Observational Study of Intestinal Flora in Infants
Brief Title: A Cohort Analysis Study of Intestinal Flora in Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mizu Jiang (Other)
Responsible Party: Sponsor-Investigator, Mizu Jiang, Director of Gastroenterology Laboratory of the Affiliated Children's Hospital of Zhejiang University Medical School, Zhejiang University
Organization: Zhejiang University (Other)
Other Study IDs: MJiang
Record Dates: First submitted 2017-12-22; First posted 2018-01-10 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Gastrointestinal Microbiome
Keywords: Gastrointestinal Microbiome; Infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Feces and human breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the influence factors of gastrointestinal microbiome in infants.

DETAILED DESCRIPTION:
The gastrointestinal microbiome is believed to be critically important for infant growth and development. As we all know, the gut microbiota can influence gut maturation, metabolic, immune and brain development in early life. Host genotype, gestational age, antibiotic use, mode of delivery, diet and the context in which the infant is born (rural vs urban, presence of siblings, pets and other factors) can influence the development of infant gut microbiota. In the early life stage, intestinal flora disorders may alter the host immune function and increase the susceptibility to immune or metabolic diseases.

This research intends to establish a birth cohort of healthy newborns. The influence factors of gastrointestinal microbiome will be investigated by means of questionnaire survey, specimen collection and high throughput sequencing analysis. What's more, the correlation of gut microbiome, infant growth as well as related diseases will be explored either. The results will provide constructive suggestions for the establishment of infant normal intestinal flora and play an indispensable role in exploring the occurrence, development and prevention of related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborns

Exclusion Criteria:

* Newborns with diseases such as congenital heart disease or congenital malformation and so on

Max Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Residents of the city of Hangzhou
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-12-22 (Actual); Primary Completion 2020-06-22 (Estimated); Study Completion 2020-12-22 (Estimated)

PRIMARY OUTCOMES:
Intestinal Flora Sequencing | Intestinal Flora Sequencing Change from Baseline to 12 months after Birth
  Intestinal Flora Sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Mizu Jiang, Doctor, Principal Investigator — The Affiliated Children's Hospital of Zhejiang University Medical School
Locations (1):
- The Gastroenterology Laboratory, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after Publication
Access Criteria: All the Researchers who Studied the Influence Factors of Intestinal Flora
URL: http://www.medresman.org

REFERENCES:
- [Background] Martin R, Makino H, Cetinyurek Yavuz A, Ben-Amor K, Roelofs M, Ishikawa E, Kubota H, Swinkels S, Sakai T, Oishi K, Kushiro A, Knol J. Early-Life Events, Including Mode of Delivery and Type of Feeding, Siblings and Gender, Shape the Developing Gut Microbiota. PLoS One. 2016 Jun 30;11(6):e0158498. doi: 10.1371/journal.pone.0158498. eCollection 2016. PMID 27362264
- [Background] Arrieta MC, Stiemsma LT, Amenyogbe N, Brown EM, Finlay B. The intestinal microbiome in early life: health and disease. Front Immunol. 2014 Sep 5;5:427. doi: 10.3389/fimmu.2014.00427. eCollection 2014. PMID 25250028
- [Background] Wopereis H, Oozeer R, Knipping K, Belzer C, Knol J. The first thousand days - intestinal microbiology of early life: establishing a symbiosis. Pediatr Allergy Immunol. 2014 Aug;25(5):428-38. doi: 10.1111/pai.12232. Epub 2014 Jun 5. PMID 24899389
- [Background] Azad MB, Konya T, Maughan H, Guttman DS, Field CJ, Chari RS, Sears MR, Becker AB, Scott JA, Kozyrskyj AL; CHILD Study Investigators. Gut microbiota of healthy Canadian infants: profiles by mode of delivery and infant diet at 4 months. CMAJ. 2013 Mar 19;185(5):385-94. doi: 10.1503/cmaj.121189. Epub 2013 Feb 11. PMID 23401405
- [Background] Penders J, Gerhold K, Stobberingh EE, Thijs C, Zimmermann K, Lau S, Hamelmann E. Establishment of the intestinal microbiota and its role for atopic dermatitis in early childhood. J Allergy Clin Immunol. 2013 Sep;132(3):601-607.e8. doi: 10.1016/j.jaci.2013.05.043. Epub 2013 Jul 27. PMID 23900058
- [Background] Penders J, Gerhold K, Thijs C, Zimmermann K, Wahn U, Lau S, Hamelmann E. New insights into the hygiene hypothesis in allergic diseases: mediation of sibling and birth mode effects by the gut microbiota. Gut Microbes. 2014 Mar-Apr;5(2):239-44. doi: 10.4161/gmic.27905. Epub 2014 Jan 23. PMID 24637604
- [Background] Backhed F, Roswall J, Peng Y, Feng Q, Jia H, Kovatcheva-Datchary P, Li Y, Xia Y, Xie H, Zhong H, Khan MT, Zhang J, Li J, Xiao L, Al-Aama J, Zhang D, Lee YS, Kotowska D, Colding C, Tremaroli V, Yin Y, Bergman S, Xu X, Madsen L, Kristiansen K, Dahlgren J, Wang J. Dynamics and Stabilization of the Human Gut Microbiome during the First Year of Life. Cell Host Microbe. 2015 Jun 10;17(6):852. doi: 10.1016/j.chom.2015.05.012. Epub 2015 Jun 10. No abstract available. PMID 26308884
- [Background] Laursen MF, Zachariassen G, Bahl MI, Bergstrom A, Host A, Michaelsen KF, Licht TR. Having older siblings is associated with gut microbiota development during early childhood. BMC Microbiol. 2015 Aug 1;15:154. doi: 10.1186/s12866-015-0477-6. PMID 26231752
- [Background] Nermes M, Endo A, Aarnio J, Salminen S, Isolauri E. Furry pets modulate gut microbiota composition in infants at risk for allergic disease. J Allergy Clin Immunol. 2015 Dec;136(6):1688-1690.e1. doi: 10.1016/j.jaci.2015.07.029. Epub 2015 Sep 3. No abstract available. PMID 26343452
- [Background] Hooper LV, Gordon JI. Commensal host-bacterial relationships in the gut. Science. 2001 May 11;292(5519):1115-8. doi: 10.1126/science.1058709. PMID 11352068
- [Background] Le Chatelier E, Nielsen T, Qin J, Prifti E, Hildebrand F, Falony G, Almeida M, Arumugam M, Batto JM, Kennedy S, Leonard P, Li J, Burgdorf K, Grarup N, Jorgensen T, Brandslund I, Nielsen HB, Juncker AS, Bertalan M, Levenez F, Pons N, Rasmussen S, Sunagawa S, Tap J, Tims S, Zoetendal EG, Brunak S, Clement K, Dore J, Kleerebezem M, Kristiansen K, Renault P, Sicheritz-Ponten T, de Vos WM, Zucker JD, Raes J, Hansen T; MetaHIT consortium; Bork P, Wang J, Ehrlich SD, Pedersen O. Richness of human gut microbiome correlates with metabolic markers. Nature. 2013 Aug 29;500(7464):541-6. doi: 10.1038/nature12506. PMID 23985870